CLINICAL TRIAL: NCT04317391
Title: Impact of Psychology on Life Quality in Chronic and Cancer Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-08-008A
Record Dates: First submitted 2020-03-17; First posted 2020-03-23 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain Syndrome; Psychology, Social
Keywords: chronic pain; Mindfulness based stress reduction; psychology; pain management program
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain management program (Experimental): All enrolled patients participate in a 20 hour pain management program over a period of 8 weeks. The program is based on Mindfulness Based Stress Reduction with modifications to fulfill needs of the Taiwanese chronic pain population.
  Interventions: Behavioral: Pain management program

INTERVENTIONS:
Behavioral: Pain management program — Mindfulness based stress reduction

SUMMARY:
This study is to compare the effect of pain management program. We compare life quality, pain scores, sleep, anxiety and depression scores, and self report measures before and after mindfulness based pain management workshops.

DETAILED DESCRIPTION:
Chronic pain is a growing problem in modern society. One in every five person in developed countries have this condition. Chronic pain is pain that persists longer than six months. It lead to psychological disorders such as anxiety, depression, anger and chronic fatigue. It decreases life quality, lower self-esteem and decrease work force. Because of these factors and the high cost of treatment, it impacts social economics highly. Chronic pain is caused by wind-up effect of the nervous system which the inhibitory signals are impaired. The nervous systems is therefore tuned up. Mindfulness based pain management helps lower this wind-up effect by noticing self, to observe and release stress. It has been proven to alter brain activity, enhance self control, improve attention and decrease secretion of stress hormones. It decreases pain and allow patients to regain control of life.

ELIGIBILITY:
Inclusion Criteria:

* Pain condition for over six months, with diagnosis by pain physician to be of chronic pain or cancer pain.

Exclusion Criteria:

* Patients unable to communicate in Mandarin.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Baseline Brief Pain inventory | Baseline
  Assesses the severity of pain and its impact on functioning
Four week Brief Pain inventory | Participants answer questionnaire at 4 weeks into pain management program
  Assesses the severity of pain and its impact on functioning
Eight weeks Brief Pain inventory | Participants answer questionnaire at 8 weeks into pain management program
  Assesses the severity of pain and its impact on functioning
One year Brief Pain inventory | Participants answer questionnaire at one year after completion of pain management program
  Assesses the severity of pain and its impact on functioning

SECONDARY OUTCOMES:
Baseline Visual analog scale | Baseline
  Pain scale at numbers 0 to 10
Four week Visual analog scale | Participants answer questionnaire at 4 weeks into pain management program
  Pain scale at numbers 0 to 10
Eight week Visual analog scale | Participants answer questionnaire at 8 weeks into pain management program
  Pain scale at numbers 0 to 10
One year Visual analog scale | Participants answer questionnaire at one year after completion of pain management program
  Pain scale at numbers 0 to 10
Baseline Pain self-efficacy questionnaire | Baseline
  Assess the confidence people with ongoing pain have in performing activities while in pain.
Four week Pain self-efficacy questionnaire | Participants answer questionnaire at 4 weeks into pain management program
  Assess the confidence people with ongoing pain have in performing activities while in pain.
Eight week Pain self-efficacy questionnaire | Participants answer questionnaire at 8 weeks into pain management program
  Assess the confidence people with ongoing pain have in performing activities while in pain.
One year Pain self-efficacy questionnaire | Participants answer questionnaire at one year after completion of pain management program
  Assess the confidence people with ongoing pain have in performing activities while in pain.
Baseline Pain catastrophizing scale | Baseline
  self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations
Four week Pain catastrophizing scale | Participants answer questionnaire at 4 weeks into pain management program
  self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations
Eight week Pain catastrophizing scale | Participants answer questionnaire at eight weeks into pain management program
  self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations
One year Pain catastrophizing scale | Participants answer questionnaire at one year after completion of pain management program
  self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations
Baseline Depression, anxiety, and positive outlook scale | Baseline
  Assess mood in pain patients
Four week Depression, anxiety, and positive outlook scale | Participants answer questionnaire at 4 weeks into pain management program
  Assess mood in pain patients
Eight week Depression, anxiety, and positive outlook scale | Participants answer questionnaire at 8 weeks into pain management program
  Assess mood in pain patients
One year Depression, anxiety, and positive outlook scale | Participants answer questionnaire at one year after completion of pain management program
  Assess mood in pain patients
Baseline Chronic Pain Acceptance Questionnaire | Baseline
  Assessment of acceptance of pain.
Four week Chronic Pain Acceptance Questionnaire | Participants answer questionnaire at 4 weeks into pain management program
  Assessment of acceptance of pain.
Eight week Chronic Pain Acceptance Questionnaire | Participants answer questionnaire at 8 weeks into pain management program
  Assessment of acceptance of pain.
One year Chronic Pain Acceptance Questionnaire | Participants answer questionnaire at one year after completion of pain management program
  Assessment of acceptance of pain.
Baseline Five Facet Mindfulness Questionnaire | Baseline
  Assessment on the five aspects of mindfulness
Four week Five Facet Mindfulness Questionnaire | Participants answer questionnaire at 4 weeks into pain management program
  Assessment on the five aspects of mindfulness
Eight week Five Facet Mindfulness Questionnaire | Participants answer questionnaire at 8 weeks into pain management program
  Assessment on the five aspects of mindfulness
One year Five Facet Mindfulness Questionnaire | Participants answer questionnaire at one year after completion of pain management program
  Assessment on the five aspects of mindfulness
Baseline Pittsburgh Sleep Quality Index | Baseline
  Assesses sleep quality
Four week Pittsburgh Sleep Quality Index | Participants answer questionnaire at four weeks into pain management program
  Assesses sleep quality
Eight week Pittsburgh Sleep Quality Index | Participants answer questionnaire at 8 weeks into pain management program
  Assesses sleep quality
One year Pittsburgh Sleep Quality Index | Participants answer questionnaire at one year after completion of pain management program
  Assesses sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided